CLINICAL TRIAL: NCT01654523
Title: Awareness Enhancement and Monitoring Device for Treatment of Trichotillomania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joseph Himle, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00050426; 2R42MH077362-02 (NIH)
Record Dates: First submitted 2012-05-10; First posted 2012-07-31 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-06

CONDITIONS: Trichotillomania
Keywords: Trichotillomania
MeSH Terms: conditions — Trichotillomania | interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Other): Open trial with no randomization
  Interventions: Device: Awareness Enhancement and Monitoring Device for Treatment of Trichotillomania

INTERVENTIONS:
Device: Awareness Enhancement and Monitoring Device for Treatment of Trichotillomania — Awareness Enhancement and Monitoring Device for Treatment of Trichotillomania
  Other Names: AEMD

SUMMARY:
The goals of the study are to further design, develop, and test an awareness enhancement and monitoring device, which will be used in the self-awareness training and general treatment of patients with compulsive hair-pulling behaviors, or trichotillomania.

DETAILED DESCRIPTION:
DESCRIPTION (provided by applicant): The goal of the proposed research is to further refine and evaluate an inconspicuous, awareness- enhancement and monitoring device (AEMD) which will assist the treatment of trichotillomania (TTM). TTM is associated with significant impairments in social functioning and often has a profound negative impact on self- esteem and well being. Conservative estimates suggest that 0.6% percent of the US population, or about 1.8 million people, meet full diagnostic criteria for TTM and approximately 7.5 million US residents have significant hair pulling problems. Of those treated, 60% to 70% are wholly or partially refractory to standard behavioral and pharmacological treatments and could therefore potentially benefit from this device. Best practice treatment for TTM involves a form of behavioral therapy known as habit reversal therapy (HRT). HRT requires persons with TTM to be aware of their hair pulling behaviors, yet the majority of persons with TTM pull most of their hair outside of their awareness. HRT also requires TTM sufferers to record the frequency and duration of their hair pulling behaviors yet it is impossible for a person to monitor behaviors that they are unaware of. Our Phase I efforts have produced a prototype device (AEMD) that solves these two problems. The prototype AEMD signals the TTM sufferer if their hand approaches their hair, thereby bringing pulling-related behavior into awareness. The prototype AEMD also logs the time, date, duration, and user classification of hair pulling related events. Our published pilot study and subsequent investigations establish that the prototype AEMD successfully alerts TTM sufferers to pulling-related behaviors and monitors TTM-related behavior in a laboratory setting. With respect to technological innovation, this project has the potential to develop the first available miniaturized, wearable, patient interactive, real-time data collecting and proximity-sensing device that both alerts sufferers to the presence of mental illness symptoms as they occur and keeps track of the frequency and intensity of the problem. The patented technologies developed for the AEMD have the potential to be of great value for a range of other health/mental health conditions or industrial applications. Our overall Phase II aim is to further refine the AEMD and to evaluate its acceptance and utility when used in an open trial course of professionally-led habit reversal therapy. It is hypothesized that the AEMD will be enthusiastically accepted by TTM sufferers and their clinicians and that it will perform as designed during the clinical trial. The Phase II AEMD will include a bracelet(s)/watch to be worn on each wrist, another element to be placed at the rear base of the neck, and a pager-like alert device to be worn at the belt-line or in a pocket. The AEMD, if found to be useful and effective, has the potential to significantly reduce the symptoms of TTM and its associated functional impairments. The AEMD also has great potential to improve assessment and monitoring of TTM behaviors which could be invaluable to clinicians planning treatment and to researchers evaluating the efficacy of various treatment strategies.

We discovered that the electronic monitoring capability of the AEMD did not function properly. Therefore we cannot report time spent pulling using the electronic device. We relied on self-report instruments to assess the impact of the psychotherapy combined with with the device on the severity of trichotillomania.

ELIGIBILITY:
Inclusion Criteria:

* Must have active hair pulling over the month prior to enrollment
* Must have noticeable hair loss
* Must experience significant distress related to Trichotillomania
* Must primarily pull from the head area
* Subjects taking medications will be included
* Must be able to read/write English

Exclusion Criteria:

* Current substance use diagnosis
* Chronic neurological disorder (other than chronic tics)
* Mental retardation
* Schizophrenia and other psychotic disorders
* Bipolar I disorder
* Prominent suicidal/homicidal ideation with imminent risk

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2005-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Himle, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 33 people were consented and interviewed for participation; 20 met study criteria and agreed to continued with the project.
Groups:
- Awareness Enhancement and Monitoring Device: Open trial with no randomization
  Awareness Enhancement and Monitoring Device for Treatment of Trichotillomania: Awareness Enhancement and Monitoring Device for Treatment of Trichotillomania
Period: Overall Study
Arm/Group | Awareness Enhancement and Monitoring Device
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.93 (9.635)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
NIMH Trichotillomania Severity and Impairment Scale [Mean (Standard Deviation); unit: units on a scale] — The NIMH Trichotillomania Severity and Impairment Scale was used to measure baseline severity and associated functional impairment of trichotillomania. This clinician-rated instrument yields a severity score that measures average time spent pulling, time spent pulling on the previous day, resistance to pulling urges, distress associated with pulling, and interference related to trichotillomania. Each item yields a score from 0 - 5 with 5 indicating the highest severity, resulting in a total of 25 possible points.
  units on a scale | 13.00 (4.04)
Massachusetts General Hospital Hair Pulling Scale [Mean (Standard Deviation); unit: units on a scale] — The Massachusetts General Hospital Hair Pulling Scale was used to measure the severity and associated functional impairment related to trichotillomania. This self-report instrument yields a total severity score. It contains seven items. Each item on this scale yields a score from 0 - 4 with 4 indicating the highest severity. The lowest possible total score is zero and the highest possible score, indicating highest severity of trichotillomania is 28.
  units on a scale | 16.12 (4.07)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Massachusetts General Hospital Hairpulling Scale Baseline to Post-treatment
Description: Measures severity of trichotillomania. Total score ranges from 0 (none) to 28 (severe). Mean change is determined by score at baseline minus score after treatment.
Time Frame: Baseline to post treatment; typically over 9 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Awareness Enhancement and Monitoring Device: Open trial with no randomization
  Awareness Enhancement and Monitoring Device for Treatment of Trichotillomania
Arm/Group | Awareness Enhancement and Monitoring Device
Number analyzed (Participants) | 19
Units on a scale | 6.695 (5.505)
Statistical Analysis 1: Comparison: Awareness Enhancement and Monitoring Device; Test type: Superiority or Other; p < 0.05, Paired t-test; Mean change in the single arm trial = 6.695, 95% CI 2-sided [4.041 to 9.348], Standard Deviation 5.505

ADVERSE EVENTS:
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes